CLINICAL TRIAL: NCT04417504
Title: Metabolic and Prolonged Satiety Effects of a Breakfast Kit: a Randomized Controlled Trial
Brief Title: Metabolic and Prolonged Satiety Effects of a Breakfast Kit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MobFood
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-11

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MobFood breakfast kit (Experimental)
  Interventions: Other: MobFood breakfast kit
- Control isocaloric breakfast (Experimental)
  Interventions: Other: Control isocaloric breakfast

INTERVENTIONS:
Other: MobFood breakfast kit — Cereal biscuit with orange fruit, cheese with fruit preparation and beverage based on oat, milk and mocha (without added sugar), specifically developed for the project MobFood_PPS4.
  Arms: MobFood breakfast kit
Other: Control isocaloric breakfast — White bread, butter and milk.
  Arms: Control isocaloric breakfast

SUMMARY:
The mobilizing programme MobFood - mobilizing scientific knoweledge and technology to answer the current nutrition market challenges - is formed by a consortium of 47 collaborative entities, between the industry and ENESIIs (Entidades Não Empresariais do Sistema de Investigação e Inovação) and is financed by Structural European Funds of Investment.

The project is currently investigating and undertaking collaborative scientific and technological strategies based on R&D and innovation, in order to boost and promote a more competitive national food industry, capable of overcoming the current challenges, including those of the Millennial Generation. This group is particularly conscious of the impact of food behaviour and food choices on health but extremely vulnerable to dietary imbalance. Strategies to improve Millenials' nutrition while providing conscious food products are needed.

This study is a randomised, cross-over controlled trial designed to test the metabolic effect, particularly in terms of appetite control and glycaemic response of a breakfast kit (nutritionally balanced and innovative), recently developed as part of the collaborative project MobFood_PPS4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Born between 1981 and 1996;
* Body mass index (BMI) between 18.5 kg/m2 and 24.9 kg/m2;
* Normoglycemic according to American Diabetes Association criteria [Fasting Plasma Glucose < 100 mg/dl, 2-h plasma glucose value during a 75 g oral glucose tolerance test (OGTT) < 140 mg/dl)];
* Healthy.

Exclusion Criteria:

* Overweight or obese (BMI ≥ 25,0 kg/m2);
* Recent body weight loss/gain >10%, within previous 3 months;
* Being on a weight loss/other special diet (e.g. Paleo diet, Atkins diet, flexitarian diet or ketogenic diet), within previous 3 months;
* Clinically significant illness, including:

type 1 or type 2 diabetes; liver disease e.g. cirrhosis; malignancy; pancreatitis or other malabsorption; gastrointestinal disorders e. g. intestinal bowel disorder, celiac disease; previous weight loss surgery e.g. bariatric surgery; chronic respiratory, neurological, psychiatric, musculoskeletal diseases/conditions; diagnosed eating disorders.

* Individuals who don't regularly consume breakfast;
* Having taken antibiotics within the 12 weeks prior to beginning the study;
* Taking other medication that could potentially affect body weight, glucose metabolism and/or appetite (e.g. GLP-1 analogues);
* Being engaged in competitive sports;
* Having >14 or >8 (males and females, respectively) alcoholic units/week; misuse of drugs;
* Having donated blood within one month prior to the beginning of the study;
* Nut or milk allergy, or other food allergy or intolerance that would compromise compliance with the study protocol;
* Pregnant or breastfeeding.

Ages: 23 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the incremental area under the curve (iAUC, mg/dl*min) for glucose response between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for glucose will be calculated based on the concentration curve following consumption of the test and control products, over 2h
Differences in the iAUC (pmol/l*min) for glucagon-like peptide-1 (GLP-1) between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for GLP-1 will be calculated based on the concentration curve following consumption of the test and control products, over 3h
Differences in the iAUC (pmol/l*min) for peptide YY (PYY) between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for PYY will be calculated based on the concentration curve following consumption of the test and control products, over 3h
Differences in the iAUC (pmol/l*min) for cholecystokinin (CKK) between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for CKK will be calculated based on the concentration curve following consumption of the test and control products, over 3h
Differences in the iAUC (pmol/l*min) for ghrelin between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for ghrelin will be calculated based on the concentration curve following consumption of test and control products, over 3h
Differences in the iAUC (pmol/l*min) for glucagon between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for glucagon will be calculated based on the concentration curve following consumption of the test and control products, over 3h

SECONDARY OUTCOMES:
Differences in the iAUC (mg/dl*min) for triacylglycerides (TG) between 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for TG will be calculated based on the concentration curve following consumption of the test and control products, over 3h
Differences in the iAUC for (mmol/l*min) non-esterified fatty acids (NEFA) between 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  The iAUC for NEFA will be calculated based on the concentration curve following consumption of the test and control products, over 3h
Differences in subjective feelings of hunger/satiety between the 2 arms | at CID1 (1 week after screening) and CID2 (at least 2 days after visit 1)
  Difference in subjective feelings of hunger/satiety from fasting state to post-prandial state with the consumption of the test and control products

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School, NOVA University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided